CLINICAL TRIAL: NCT00624949
Title: Aortic Dimensions, 24hour Ambulatory Blood Pressure and Sympathovagal Tone in Turner Syndrome. In Relation to Aortic Dilatation and Dissection.
Brief Title: Aortic Dimensions in Turner Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Professor Jens Sandahl Christiansen, Aarhus University Hospital, Aarhus, Denmark
Other Study IDs: 20010248
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Turner Syndrome
Keywords: Turner syndrome; aortic dimensions; blood pressure; aortic dilatation; aortic rupture
MeSH Terms: conditions — Turner Syndrome; Aortic Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: women with Turner syndrome
- 2.: Control women

SUMMARY:
An observational study of 102 women with Turner syndrome followed for 6 years with a two-yearly examination including ECHO, MRI of the heart and 24 ambulatory blood pressure. It has been found that besides an significantly increased risk of congenital cardiac malformations, TS have an increased risk of developing cardiac disease including the life threatening condition of aortic dilatation and rupture. The aim of the study is to describe the cardiac conditions of TS, evaluate different methods of examination and identify possible risc factors.

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome
* Age 18-70 years

Exclusion Criteria:

* Extreme adipositas
* Contraindications to a MRI scan
* Malignant disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recrutted from hospital clinics and through the patient organisation
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2003-08; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Aortic diameter at 3 well-defined levels measured by MRI and ECHO | 2-yearly for 6 years

SECONDARY OUTCOMES:
24hour ambulatory blood pressure | 24h 2-yearly for 6 years

REFERENCES:
- [Derived] Viuff M, Skakkebaek A, Johannsen EB, Chang S, Pedersen SB, Lauritsen KM, Pedersen MGB, Trolle C, Just J, Gravholt CH. X chromosome dosage and the genetic impact across human tissues. Genome Med. 2023 Mar 28;15(1):21. doi: 10.1186/s13073-023-01169-4. PMID 36978128
- [Derived] Trolle C, Mortensen KH, Bjerre M, Hougaard DM, Cohen A, Andersen NH, Gravholt CH. Osteoprotegerin in Turner syndrome - relationship to aortic diameter. Clin Endocrinol (Oxf). 2015 Mar;82(3):397-403. doi: 10.1111/cen.12522. Epub 2014 Jul 2. PMID 24923356
- [Derived] Trolle C, Mortensen KH, Pedersen LN, Berglund A, Jensen HK, Andersen NH, Gravholt CH. Long QT interval in Turner syndrome--a high prevalence of LQTS gene mutations. PLoS One. 2013 Jul 25;8(7):e69614. doi: 10.1371/journal.pone.0069614. Print 2013. PMID 23936059